CLINICAL TRIAL: NCT07380386
Title: A Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SKB105 for Injection in Participants With Advanced Solid Tumors
Brief Title: SKB105 for Injection in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB105-I/II-01
Record Dates: First submitted 2026-01-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: SKB105; Integrin β6 (ITGB6)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB105 monotherapy (Experimental): Subject will be dosed with SKB105 for injection every 3 weeks(q3w)
  Interventions: Drug: SKB105 for injection Monotherapy

INTERVENTIONS:
Drug: SKB105 for injection Monotherapy — SKB105 for injection monotherapy, iv drip, every 3 weeks (Q3W), until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.
  Other Names: SKB105 Antibody-Drug Conjugate(ADC) in solid tumors

SUMMARY:
This is a Phase 1/2 clinical study to evaluate the safety and efficacy of SKB105 in participants with advanced solid tumors. The study includes a dose escalation stage, a dose expansion stage, and a indication expansion stage.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1/2 clinical study to evaluate the safety, tolerability, Pharmacokinetics(PK) characteristics, immunogenicity, and efficacy of SKB105 in participants with advanced solid tumors. The study includes a Phase 1 dose escalation stage, a Phase 1 dose expansion stage, and a Phase 2 indication expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily joined this study and signed an informed consent form.
2. The age at the time of signing the informed consent form must be between 18 and 75 years.
3. Participants with histologically or cytologically confirmed advanced solid tumors who have failed standard therapy, have no standard therapy available, or are intolerant to standard therapy.
4. Participants should provide tumor tissue samples for biomarker testing as much as possible during the screening period;
5. Researchers evaluated based on Response Evaluation Criteria in Solid Tumors(RECIST) Version 1.1 that there is at least one measurable lesion present.
6. Eastern Cooperative Oncology Group (ECOG) score is 0 or 1.
7. Expected survival period ≥ 12 weeks.
8. Participants have sufficient bone marrow, liver, kidney, and coagulation functions.
9. Male and female participants must agree to use highly effective contraceptive methods during the study period.

Exclusion Criteria:

1. Participants known to have meningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, and active central nervous system (CNS) metastasis.
2. Patients with other malignant tumors within 3 years before the first administration.
3. There are serious heart or vascular diseases or high-risk factors present.
4. According to researchers' judgment, it is an uncontrollable systemic disease.
5. There are pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage (>1 time/week).
6. History of interstitial lung disease or non infectious pneumonia.
7. There are other lung diseases that may interfere with drug-related pulmonary toxicity.
8. Severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or a history of corneal diseases that hinder/delay corneal healing.
9. The toxicity of previous anti-tumor treatments has not been relieved, defined as the toxicity has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Version 6.0 grade 0 or 1.
10. There is a risk of developing esophagotracheal fistula or esophageal pleural fistula, or tumor invasion or compression of surrounding important organs and blood vessels accompanied by related clinical symptoms.
11. Within 3 months prior to the first administration, there have been clinical symptoms of intestinal obstruction, gastrointestinal perforation or fistula, urethral fistula, and abdominal abscess.
12. Serious infection occurred within 4 weeks before the first administration.
13. Active hepatitis B or C, or simultaneous infection with Hepatitis B virus(HBV) and Hepatitis C virus(HCV).
14. Human immunodeficiency virus (HIV) test is positive or there is a history of acquired immunodeficiency syndrome (AIDS); Known active syphilis infection.
15. Known active pulmonary tuberculosis.
16. Known history of allogeneic organ transplantation or hematopoietic stem cell transplantation.
17. History of allergies to any components of SKB105 injection or severe hypersensitivity reactions to other monoclonal antibodies.
18. Previously received drug therapy targeting Integrin β6(ITGB6) or any form of drug therapy containing topoisomerase I inhibitors.
19. Received chemotherapy, immunotherapy, biological therapy, or other large molecule anti-tumor drugs within 4 weeks before the first administration;
20. Within 6 months prior to the first administration, lung lesions received radiation therapy with a total dose greater than 30 Gray.
21. Have undergone major surgical procedures or suffered serious injuries within 28 days prior to the first administration of medication.
22. Those who have received treatment with other clinical investigational drugs within 28 days prior to their first administration.
23. Individuals who have previously received anti-tumor vaccines or have received any active vaccines within 28 days prior to their first treatment with the investigational drug.
24. Participants who received systemic corticosteroid therapy or other immunosuppressive drugs with>10 mg/day prednisone within 2 weeks prior to the first dose.
25. Within 14 days before the first administration or within 5 half lives of known drugs (whichever is longer), she received a strong inhibitor or strong inducer of cytochrome P450 or a breast cancer resistance protein (BCRP) inhibitor.
26. Pregnant or lactating women.
27. Participants with a known history of mental illness or substance abuse are unable to cooperate in completing the study.
28. Suffering from local or systemic diseases caused by non malignant tumors, or diseases or symptoms secondary to tumors, which may affect compliance.
29. Any condition that the researcher deems to interfere with the evaluation of the investigational drug, the safety of participants, or the interpretation of research results, or any other condition that the researcher deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From date of initial dose until up to 21 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during first 21 days and is at least possibly related to study drug.
Objective Response Rate (ORR) | up to 3 years
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 3 years
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 3 years
  Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Jin, Study Director
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shangahi Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No